CLINICAL TRIAL: NCT00205335
Title: The Impact of Increased Availability of Test Strips on Blood Glucose Control in Patients With Diabetes
Brief Title: Free Test Strips and Blood Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: M-2004-1069
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- glucose monitoring (Other): Each participant received a Bayer Breeze Monitor and glucose test strips for monitoring blood sugar.
  Interventions: Device: Ascencia Breeze Glucose meter; Device: Breeze Glucose Monitor (Bayer)

INTERVENTIONS:
Device: Ascencia Breeze Glucose meter — All study participants received glucose meter and test strips.
  Other Names: Ascencia Breeze glucose meters made by Bayer and test strips
Device: Breeze Glucose Monitor (Bayer) — Each participant received a Breeze monitor and glucose test strips.
  Other Names: Ascencia Breeze Glucose Meter, Bayer

SUMMARY:
This study is designed to determine if there is an impact on blood glucose control in patients who receive free test strips. Patients in the study have no insurance or insurance that does not cover the purchase of test strips. A comparison of weight, blood pressure, and Hemoglobin A1C from entry to the final visit will be used to compare patients' management of their diabetes. Recommended values for these parameters will be used as the standard for comparisons. The investigators anticipate that patients receiving free test strips will show an improvement in the listed parameters as well as in satisfaction with their care.

DETAILED DESCRIPTION:
According to the National Institutes of Diabetes and Digestive and Kidney Diseases, an estimated 16 million people in the United States have diabetes mellitus. About one third of these people don't know they have diabetes and are therefore, not receiving treatment. Another 798,000 people are diagnosed with diabetes each year.

Diabetes is the fourth leading cause of death in Wisconsin, as stated at the Wisconsin Department of Health and Family Services website. Diabetes costs an estimated annual $2.1 billion in health care costs and lost productivity. Each year, over 3,600 Wisconsin residents die from diabetes. Others experience disabling complications, including blindness, amputations, heart and kidney disease. In 1998, in Dane County alone, the direct costs of diabetes were estimated at $82.0 million and indirect costs at $100.4 million.

Two landmark studies in the United States and the United Kingdom proved that the level of blood sugar control predicts the onset and severity of diabetes-related complications for both Type 1 and Type 2 diabetes. Thus, people who are able to keep their blood sugars as close to normal as possible can reduce their risks of complications and live relatively "normal" lives. Moreover, the costs to the community will also be reduced.

In order to do this, persons with diabetes need to test blood sugar levels multiple times per day. There are a variety of meters available for testing. Many people have insurance that covers the cost of the meters and related test strips. For those who do not have this coverage, meters are often available free of charge. Unfortunately, this is not true of the test strips, which average $1 each. A person testing four times a day, seven days a week would need almost $1470 to purchase strips for a year.

In the past year, the investigators have seen 35 patients followed in either the East or West Diabetes Clinics who do not have insurance and thus, no way to pay for test strips. It can be assumed that without an adequate number of test strips, these patients are not getting the necessary information to achieve optimal blood sugar control. This puts them at risk for more complications of their diabetes with concurrent emotional and financial costs to them and their families. Further, the cost to the community in the long run is increased.

2. Describe the design of your study. Use care to distinguish experimental interventions from standard medical treatment. Specifically include the following information:

The investigators will enroll 35 subjects identified in either the East or West diabetes clinic who do not have insurance or who are underinsured. Underinsured indicates patients with insurance that does not cover the purchase of test strips. Certified Diabetes Educators (CDE) identified other patients after an initial visit when lack of adequate insurance coverage was noted. The list of identified patients was sent to the patient's physician and CDE. Two patients were eliminated who are self-pay by choice; they are self-employed and have adequate resources. Other subjects were eliminated for the following criteria: discharge from UWHC Diabetes Clinic to a primary care provider; patients whose diabetes is controlled by diet alone; patients who are incarcerated and currently have coverage through the penal system.

Subjects will be provided a voucher to obtain free test strips. Subjects routinely return to the clinic at 4-month intervals (study entry, months 4,8,12). During these visits subjects will undergo a Hemoglobin A1C, check height, weight, and blood pressure and complete satisfaction questionnaires at study entry and month 12. Only the questionnaires would not be considered standard of care.

3. What method(s) will you use to recruit subjects? Will these methods involve material inducements? Subjects who meet the eligibility criteria will be offered participation. Subjects will receive testing strips, clinic visits at entry and at months 4,8 and 12 and Hemoglobin A1C (HA1C) testing at the above intervals free of charge.

4. Does your study have a statistical justification for its sample size? For the analysis of its results? If you answer "yes" to these questions, briefly describe each justification.

No

C. Identify the potential risks to subjects of participation in your study. Describe the expected frequency, severity, and reversibility of the major risks you identify. Include possible late effects of participation (e.g., secondary cancers).

All subject records will be kept strictly confidential according to HIPPA privacy rules. Subject records will contain only a study number. The key to the study numbering will be kept in a locked filing cabinet. Subjects may experience slight pain and bruising from the blood draws of the HA1C.

D. Identify the expected benefits to subjects of participation in your study. Also identify any potential scientific benefits produced by your study.

Subjects will receive free testing strips and free HA1C testing for a year. Subjects may experience better control of their diabetes as a result of testing their blood sugar levels.

E. Describe the procedure for obtaining the consent of each subject or the subject's parent or representative. Confirm that you have attached a copy of each consent form. The form should include all the elements of consent listed in the HSC Guidelines.

Subjects will be given the informed consent and allowed ample time to read the informed consent or have it read to them. Once the consent form has been read subjects will have as much time as needed to ask any questions they may have. Once the subject has had all of their questions answered and agrees to participate the subject will sign the consent form in the presence of the PI or a delegate. Subjects will be given a copy of the signed consent form for their records.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of diabetes who have no health insurance or insurance that does not pay for purchase of blood test strips

Exclusion Criteria:

* Patients with a diagnosis of diabetes who have health insurance that pays for purchase of blood test strips

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Weight | one year
Blood pressure | one year
Hemoglobin A1C | one year

SECONDARY OUTCOMES:
Satisfaction with care | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sherree Drezner, ACSW, LCSW, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States